CLINICAL TRIAL: NCT00497809
Title: An Open-Label, Dose Finding, Prospective, Multi Center, Randomized, Parallel Group Study to Assess the Efficacy and Safety of Three Different Dose Levels of AVI 014 (G-CSF) Compared With a Standard Dose of Neupogen® in Breast Cancer Patients at High (>20%) Risk for Chemotherapy Induced Severe Neutropenia
Brief Title: Safety and Efficacy Study of GCSF Therapy to Treat Patients at High Risk for Chemotherapy Induced Severe Neutropenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AviGenics (Industry)
Responsible Party: Mark Hites, Director, Regulatory Affairs, AviGenics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVI-014-P02
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer; Neutropenia
Keywords: Breast Cancer; Neutropenia; Chemotherapy; High risk
MeSH Terms: conditions — Breast Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): AVI-014 2.5mcg/kg
  Interventions: Drug: AVI-014 versus Filgrastim
- 2 (Experimental): AVI-014 5.0 mcg/kg
  Interventions: Drug: AVI-014 versus Filgrastim
- 3 (Experimental): AVI014 10.0 mcg/kg
  Interventions: Drug: AVI-014 versus Filgrastim
- 4 (Active Comparator): Filgrastim 5.0 mcg/kg
  Interventions: Drug: AVI-014 versus Filgrastim

INTERVENTIONS:
Drug: AVI-014 versus Filgrastim — 3 different dose arms of AVI-014 versus Filgrastim for up to 14 days daily

SUMMARY:
The overall purpose of this study is to assess the dose response, efficacy, and safety of three different dose levels of AVI 014 (granulocyte colony-stimulating factor [G-CSF]) in breast cancer patients at high (>20%) risk for chemotherapy-induced severe neutropenia.

DETAILED DESCRIPTION:
Filgrastim is a recombinant human G-CSF (rhG-CSF) developed in the mid 1980s, and was approved by the United States (US) Food and Drug Administration (FDA) for use in chemotherapy induced neutropenia in 1991 under the trade name Neupogen®. Filgrastim was first approved in the EU in Germany in 2001 under the same trade name. Filgrastim is a non glycosylated protein, produced in E. coli bacteria transfected with rhG-CSF copy deoxyribonucleic acid (cDNA). Filgrastim differs from native human G CSF only in the addition of an N terminal methionine required for expression in a bacterial host. In 2002, a pegylated filgrastim with extended duration of action relative to the naked filgrastim was approved by the FDA and the EU Commission under the trade name Neulasta.

AviGenics has generated transgenic hens carrying rhG CSF cDNA, which express a glycosylated form of rhG-CSF protein in their egg white. The purified rhG-CSF is biologically active, as assessed by its in vitro binding and cell proliferation activities, and has been fully characterized by AviGenics. AviGenics intends to develop this product to treat chemotherapy-induced neutropenia.

The overall goal of this study is to assess dose response, efficacy, and safety of three different dose levels of AVI-014 (G-CSF) in breast cancer patients at high (>20%) risk for chemotherapy induced severe neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily provide written informed consent before screening, following an explanation of the nature and purpose of this study.
* Women, aged 18 years and older
* Histologically confirmed breast cancer, undergoing one of a variety of chemotherapy regimens, or with other risk factors that could lead to a >20% risk of developing severe neutropenia. Patients receiving chemotherapy regimens with high-risk for severe neutropenia are eligible; eligibility of patients receiving intermediate-risk chemotherapy regimens must be discussed with the Medical Monitor for the presence of additional patient-specific risk factors.
* Must be receiving first-line adjuvant or neoadjuvant therapy for localized breast cancer or first-line chemotherapy for metastatic breast cancer. It is recommended that patients with human epidermal growth factor receptor 2 (HER2/neu)-positive breast cancer should be receiving Herceptin® (trastuzumab), if approved and available for this indication.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of grade 0 to 2
* Adequate renal (serum creatinine and blood urea nitrogen [BUN] <3 times the upper limit of normal [ULN]) and hepatic (serum bilirubin, aspartate aminotransferase [AST], and alanine aminotransferase [ALT] <3 times ULN) function.
* Able to adhere to the study visit schedule and other protocol requirements.
* Women who are not pregnant and do not plan to become pregnant during the study. Women of childbearing potential must have a negative serum pregnancy test result within seven days before the first dose of study drug and must be using adequate non hormonal barrier contraception before entering the study and throughout the study. Non childbearing potential is defined as post-menopausal for at least one year, surgically sterile, or having had a hysterectomy before study start.

Exclusion Criteria:

* Pregnant or lactating women.
* History or clinical evidence of a serious medical illness, including renal, hepatic, respiratory, cardiovascular, endocrine, neurologic, psychiatric, or hematologic disease, which in the opinion of the investigator will interfere with study participation.
* Metastatic brain or meningeal tumors.
* Ascites or pleural effusions.
* Any active infection requiring systemic antimicrobial therapy.
* Known to be positive for human immunodeficiency virus (HIV, anti-HIV+), hepatitis B antigen (HBAg[+]), or hepatitis C antibody (HCVAb[+]).
* Known or suspected hypersensitivity to the study drug or its components, such as avian products, including influenza vaccine, or to E. coli-derived proteins.
* Currently receiving radiation therapy for treatment of a malignant condition, or have completed radiation therapy within 14 days before study entry. Radiation therapy for oncologic emergency is allowed.
* Participated in another therapeutic clinical study (i.e., not an epidemiological study or genomic screening study) during the past 30 days, or are likely to simultaneously participate in another therapeutic clinical study.
* History of, or known current problems with, substance abuse, or any medical, psychological, and/or social condition that may interfere with the patient's participation in the study, or with evaluation of the study results.
* Any condition that could jeopardize the patient's safety and compliance, as judged by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is duration of grade 4 neutropenia (DSN), defined as ANC <0.5 x 109/L during chemotherapy cycle 1. | First cycle of GCSF

SECONDARY OUTCOMES:
• Incidence of grade 4 neutropenia • Duration of neutropenia (defined as the number of days with ANC <0.5 x 109/L and <0.1 x 109/L) | Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Howard Ozer, MD, Principal Investigator — University of Oklahoma; Robert J. Grieve, M.B,Ch.B., FRCR, Principal Investigator — University Hospitals of Coventry and Warwickshire; Walter Kraft, MD, MS, FACP, Study Chair — AviGenics
Locations (31):
- United States (14):
  - Pacific Cancer Medical Center, Anaheim, California
  - California Cancer Center, Greenbrae, California
  - Ghassan Al-Jazayrly, MD, Inc., Los Angeles, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Brian LeBerthon, MD, A Medical Corporation, West Covina, California
  - Infosphere Clinical Research, West Hills, California
  - Physicians Research Alliance LLC., DeBary, Florida
  - Southern Illinois Hematology/Oncology, Centralia, Illinois
  - Gabrail Cancer Center, Canton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - University of Oklahoma Health Sciences Ctr, Oklaoma City, Oklahoma
  - Cancer Care Institute of Carolina, Aiken, South Carolina
  - Cancer Specialists of South Texas, Corpus Christi, Texas
  - Cancer Outreach Associates PC, Abingdon, Virginia
- India (17):
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Idgah Hills, Bhopal
  - Apollo Specialty Hospital, Padma Complex, 320 Mount Road, Chennai
  - Amrita Institute of Medical Sciences, Amrita Lane Elamakkara, Cochin
  - Apollo Hospitals Educational and Research Foundation, Jubilee Hills, Hyderabad
  - Kidwai Memorial Institute of Oncology, Dr. M.H. Marigowda Road, Bangalore, Karnataka
  - Mohan Dai Oswal Cancer Treatment & Research Foundation, G.T. Road, Sherpur Bye Pass, Ludhiana
  - Dayanand Medical College and Hospital, Tagore Nagar, Civil Lines, Ludhiana
  - Meenakshi Mission Hospital and Research Centre, Lake Area, Melur Road, Madurai,
  - Kasturba Medical College Hospital, Attavar, Mangalore
  - Tata Memorial Hospital,, Dr. E Borges Road, Parel, Mumbai
  - Dharamshila Hospital and research Centre, Vasundhara Enclave, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, Delhi Mathura Road, Sarita Vihar, New Delhi
  - IRCH, AIIMS, Ansari Nagar,, New Delhi, New Delhi
  - Dharamshila Cancer Center, Dharamshila Marg, Vasundhara Enclave, New Delhi
  - Regional Cancer Centre, IGIMS, Sheikhpura, Patna
  - Ruby Hall Clinic, 40 Sasoon Road, Pune
  - King George Hospital, Vizag, Vishakhapattanam